CLINICAL TRIAL: NCT06267963
Title: A PHASE 1, OPEN-LABEL, PARALLEL-GROUP, SINGLE-DOSE STUDY IN HEALTHY ADULT MALE PARTICIPANTS TO INVESTIGATE THE ABSORPTION, DISTRIBUTION, METABOLISM AND EXCRETION OF [14C]-PF-07220060 AND TO ASSESS THE ABSOLUTE BIOAVAILABILITY AND FRACTION ABSORBED OF PF-07220060 USING A 14C-MICROTRACER APPROACH
Brief Title: A Study to Understand What the Body Does to the Study Medicine Called PF-07220060 When Taken by Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C4391010; 2023-507074-40-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-01-17; First posted 2024-02-20 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Healthy Participants
Keywords: Absorption; Distribution; Metabolism; Elimination; ADME (Absorption, Distribution, Metabolism and Excretion); Pharmacokinetics; Bioavailability; Fraction absorbed; Mass balance; Healthy Males; Cyclin-Dependent Kinase 4 (CDK4) inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants will receive one dose of [14C] PF-07220060 by mouth
  Interventions: Drug: Oral [14C]PF-07220060
- Cohort 2 (Experimental): Participants will take one dose of PF-07220060 by mouth and one dose as an IV (intravenous) infusion of [14C] PF-07220060.
  Interventions: Drug: Oral PF-07220060; Drug: IV [14C] PF-07220060

INTERVENTIONS:
Drug: Oral [14C]PF-07220060 — A single oral dose of [14C]PF-07220060, will be administered as a liquid formulation in Cohort 1.
  Arms: Cohort 1
Drug: Oral PF-07220060 — A single oral dose of PF-07220060, will be administered as a liquid formulation in Cohort 2.
  Arms: Cohort 2
Drug: IV [14C] PF-07220060 — A single IV infusion of [14C]PF-07220060 will be administered in Cohort 2 at Tmax after the administration of the unlabeled oral dose.
  Arms: Cohort 2

SUMMARY:
The purpose of this study is to learn about how much PF-07220060 will be taken up and processed by healthy male participants.

The study is seeking for participants who:

* are males aged 18 to 65 years and are healthy.
* have Body mass index (BMI) between 17.5 and 30.5 kilograms/meter2
* have a total body weight of at least 50 kilograms.

The study consists of two groups. In group 1, participants will take one amount of PF-07220060 by mouth. In group 2, participants will take one amount by mouth and one amount as an injection through a vein at the study clinic.

In group 1, participants will stay at the clinic site for up to 15 days. In group 2, the duration of participants' stay depends on the results of group 1.

During their stays, participants will have their blood, urine, and feces collected by the study doctors several times. We will measure the level of PF-07220060 in participants' blood, urine, and feces samples. This will help to know how much the study medicine is getting taken up by the body. At the end of the study, participants will be contacted by phone to check in. Participants will be involved in this study for about 9 weeks from the screening until the follow-up.

ELIGIBILITY:
Key Eligibility criteria for this study include, but are not limited to the following:

Inclusion Criteria:

* Male participants aged 18 to 65 years at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body mass index (BMI) of 17.5-30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

Exclusion Criteria:

* Participants with a history of irregular bowel movements (eg, regular episodes of diarrhea or constipation, irritable bowel syndrome [IBS] or lactose intolerance).
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives (whichever is longer) preceding the first dose of study intervention used in this study. Previous exposure to PF-07220060 or participation in studies requiring PF-07220060 administration.
* Total 14C radioactivity measured in plasma exceeding 11 mBq/mL.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Cumulative recovery (%) of radioactivity in urine and feces (adjusted for vomitus, if any), expressed as a percent of total oral radioactive dose administered. | Cohort 1 pre-dose to maximum Day 14
  To characterize the rate and extent of excretion of total radioactivity following administration of a single oral dose of [14C]PF-07220060.
Amount of metabolites of [14C]PF-07220060 in plasma, urine, and feces. | Cohort 1 pre-dose to maximum Day 14
  To characterize the metabolic profile for PF- 07220060 and identify the circulating and excreted metabolites of PF-07220060 following administration of a single oral dose of [14C]PF-07220060.

SECONDARY OUTCOMES:
Dose normalized AUCinf of intravenous radiolabeled PF-07220060 in plasma (if data permit) | Cohort 2 pre-dose to maximum Day 14
  Dose normalized area under the plasma concentration-time profile from time zero extrapolated to infinite time following administration of a single intravenous dose of radiolabeled PF-07220060.
The absolute oral bioavailability (F) of PF-07220060 | Cohort 2 pre-dose to maximum Day 14
  The ratio of dose-normalized plasma AUCinf of oral PF-07220060 and IV [14C]PF-07220060
The fraction of PF-07220060 dose absorbed (Fa) | Cohort 1 predose to maximum Day 14; Cohort 2 pre-IV dose to maximum Day 14
  Fa calculated from the ratio of total recovered radioactivity [14C] in urine following single dose administration of [14C]PF-07220060 orally in Cohort
  1 and via IV infusion in Cohort 2.
Number of participants with treatment emergent clinically significant laboratory abnormalities | Both cohorts from pre-dose to 28 days post-dose
Number of participants with treatment emergent clinically significant abnormal ECG measurements | Both cohorts from pre-dose to 28 days post-dose
Number of participants with treatment emergent clinically significant abnormal vital measurements | Both cohorts from pre-dose to 28 days post-dose
Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) | Both cohorts from pre-dose to 28 days post-dose
Number of participants with treatment emergent clinically significant abnormal physical examination | Both cohorts from pre-dose to 28 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4391010